CLINICAL TRIAL: NCT01298908
Title: The Utility of Novel Ambulatory Treatment Techniques in Venous Insufficiency
Brief Title: Comparison of Treatments in Venous Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0 - Sep 6th, 2006
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Venous Insufficiency
Keywords: varicose veins, oedema
MeSH Terms: conditions — Venous Insufficiency; Varicose Veins; Edema | interventions — Laser Therapy; Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Operative treatment (Other): vein stripping
  Interventions: Procedure: Operative treatment
- Laser ablation (Other): Ultrasound guided laser ablation
  Interventions: Procedure: Laser ablation
- Foam sclerotherapy (Other): Ultrasound guided foam sclerotherapy
  Interventions: Procedure: Foam sclerotherapy

INTERVENTIONS:
Procedure: Operative treatment — In operative treatment the great saphenous vein will be removed after flush ligation by femoral vein and stripping of the trunk.
  Other Names: Vein stripping
  Arms: Operative treatment
Procedure: Laser ablation — In intravenous laser treatment a thin laser fiber is inserted through a tiny distal entry point. The probe is guided into place using ultrasound and the procedure is performed under local tumescence anesthesia. Laser energy is delivered to seal the faulty vein.
  Other Names: Ultrasound guided laser ablation
  Arms: Laser ablation
Procedure: Foam sclerotherapy — Ultrasound guided foam sclerotherapy involves an injection of foam (sodium tetradecyl sulfate mixed with air according to the Thessari method) directly into the venous trunk under ultrasound control.
  Other Names: Ultrasound guided foam sclerotherapy
  Arms: Foam sclerotherapy

SUMMARY:
Randomized controlled trial, a method used to implement the random allocation sequence is numbered containers.

The aim of the study is to compare operative treatment, ultrasound guided laser ablation and ultrasound guided foam sclerotherapy in occluding/ablating of insufficiency in great saphenous trunks. On the grounds of the available data, the study hypothesis is that using laser or operative treatment more than 20 percent better outcome can be achieved compared to foam sclerotherapy.

DETAILED DESCRIPTION:
In operative treatment the great saphenous vein will be removed after flush ligation by femoral vein and stripping of the trunk. In intravenous laser treatment a thin laser fiber is inserted through a tiny distal entry point. The probe is guided into place using ultrasound and the procedure is performed under local tumescence anesthesia. Laser energy is delivered to seal the faulty vein. Ultrasound guided foam sclerotherapy involves an injection of foam (sodium tetradecyl sulfate mixed with air according to the Thessari method) directly into the venous trunk under ultrasound control. In each group patients will use supportive treatment stockings 2 weeks after treatment. The patients in all groups are followed up one year by ultrasound scanning.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic superficial vein insufficiency
* patient must be 20-70 years old
* degree of difficulty of vein insufficiency C2-C4
* average diameter of refluxing great saphenous vein 4 -10 mm
* patient is agreeable to the study

Exclusion Criteria:

* peripheral atherosclerotic occlusive disease
* lymphoedema
* severe concomitant disease
* venous ulcers or unclassified skin changes
* BMI more than 40
* pregnancy
* allergy to the foam used in sclerotherapy or to local anaesthetics
* coagulation disorder
* bilateral vein insufficiency (equal symptoms)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recanalization or reflux of the treated venous trunk | at 1 and 12 months
  Results will be verified by Duplex scanning

SECONDARY OUTCOMES:
Symptom relief | at 1 and 12 months
  Symptoms will be evaluated by using CEAP-classification and degree of disability
Complications related to procedure | at 1 and 12 months
  At 1 month follow-up immediate complications will be recorded. At 12 months follow-up appearance of late complications and pain and incapacity for work due to the procedure will be recorded.
Quality of life | at 1 and 12 months
  Quality of life is evaluated with two questionnaires: Aberdeen (which is a 13-item questionnaire with categories related specially to disadvantages caused by varicose veins) and 15D (a questionnaire with categories related to general quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Maarit Venermo, MD,PhD, Study Director — Department of Vascular Surgery, Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Department of Vascular Surgery, Helsinki University Central Hospital, Helsinki, HUS
  - Department of Vascular Surgery, Tampere University Hospital, Tampere

REFERENCES:
- [Derived] Vahaaho S, Halmesmaki K, Alback A, Saarinen E, Venermo M. Five-year follow-up of a randomized clinical trial comparing open surgery, foam sclerotherapy and endovenous laser ablation for great saphenous varicose veins. Br J Surg. 2018 May;105(6):686-691. doi: 10.1002/bjs.10757. PMID 29652086